CLINICAL TRIAL: NCT06897592
Title: The Effect of Enneagram Training on Midwifery Students Communication, Self-confidence and Emotional Intelligence Levels: Randomized Controlled Trial
Brief Title: The Effect of Enneagram on Midwifery Students Communication, Self-confidence and Emotional Intelligence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ebru Ertas, Lecturer, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KutahyaHSU2025
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Enneagram
Keywords: communication; self-confidence; emotional intelligence
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: A randomized study with an application and a control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Experimental): Students in the application group will receive enneagram training for 2 hours once a week for 8 weeks.
  Interventions: Behavioral: Enneagram
- Control Group (No Intervention): No intervention will be applied to students in the control group.

INTERVENTIONS:
Behavioral: Enneagram — The training will be offered to students as 10 modules, 2 hours per week, for 8 weeks. The training content will consist of the Enneagram basic level and relationships.
  Arms: Training Group

SUMMARY:
This research was planned to evaluate the effects of Enneagram training on the communication skills, self-confidence and emotional intelligence levels of midwifery students. In this study, planned as a quasi-experimental randomized controlled research, with pre-test-post-retention(permanence) test will be used. Enneagram training will last 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Midwifery department 2nd-3rd-4th grade student.

Exclusion Criteria:

* Having experienced an acute traumatic event (loss of parents, divorce, accident, etc.),
* Having a psychological disorder,
* Having received training on Temperament or Enneagram.
* Requesting to withdraw from the study at any stage of the study,
* Not attending more than one training session.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 168 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The effect of 8-week Enneagram training on students communication skills | The training will last 8 weeks. At the end of the training, the final test of the Health Professionals Communication Skills Scale was administered.
  Health Professionals Communication Skills Scale will be used to evaluate communication skills of students before the training.
The effect of 8-week Enneagram training on students Self-Confidence. | The training will last 8 weeks. At the end of the training, the final test of the Self-Confidence Scale was administered.
  A self-confidence scale will be used to assess students' self-confidence before the training. The highest score that can be obtained from the scale is 165, and the lowest score is 33.
The effect of 8-week Enneagram training on students emotional intelligence trait | The training will last 8 weeks. At the end of the training, the final test of the Emotional Intelligence Trait Scale was administered.
  Emotional Intelligence Trait Scale will be used to evaluate emotional intelligence trait of students before the training.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Ertaş, Msc., Principal Investigator — Kutahya Health Sciences University; Nebahat Özerdoğan, Prof., Study Director — Eskisehir Osmangazi University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)